CLINICAL TRIAL: NCT06655311
Title: Multiple-Rising Dose Clinical Study to Evaluate the Safety and Pharmacokinetics of MK-0616 in Healthy Participants and in Male and Female Participants Taking Statins
Brief Title: A Study of Enlicitide Chloride (MK-0616) in Healthy Participants and Participants Taking Statins (MK-0616-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0616-012; MK-0616-012 (Other: MSD)
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — MK-0616

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enlicitide Chloride (Experimental): Participants receive enlicitide chloride titrated orally from Dose 1, Dose 2, or Dose 3 once daily (QD) over the course of a 14-day treatment for each dose based on the safety and tolerability of the previous starting dose. The total treatment duration is up to approximately 6 weeks.
  Interventions: Biological: Enlicitide Chloride
- Placebo (Placebo Comparator): Participants receive placebo orally for up to approximately 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Enlicitide Chloride — Oral administration
  Other Names: MK-0616
  Arms: Enlicitide Chloride
Other: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The goal of this study is to learn what happens to different doses of enlicitide chloride over time in the body of healthy participants and participants taking statins, a group of medicines used to reduce the levels of high cholesterol in the bloodstream. The researchers want to learn about the safety of enlicitide chloride when administered at high doses.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health based on medical history, physical examination, vital signs (VS) measurements, electrocardiograms (ECGs), and laboratory safety tests performed before randomization
* Has a body mass index (BMI)≥18 and ≤32 kg/m^2

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 56 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 42 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Curve from Time 0 to 24 Hours (AUC0-24) of Enlicitide Chloride | At designated timepoints (up to approximately 24 hours)
  Blood samples will be collected to determine the AUC0-24 of enlicitide chloride.
Maximum Plasma Concentration (Cmax) of Enlicitide Chloride | At designated timepoints (up to approximately 1 week)
  Blood samples will be collected to determine the Cmax of enlicitide chloride.
Plasma Concentration 24 Hours Postdose (C24) of Enlicitide Chloride | At designated timepoints (up to approximately 1 week)
  Blood samples will be collected to determine the C24 of enlicitide chloride.
Time to Maximum Plasma Concentration (Tmax) of Enlicitide Chloride | At designated timepoints (up to approximately 1 week)
  Blood samples will be collected to determine the Tmax of enlicitide chloride.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Enlicitide Chloride | At designated timepoints (up to approximately 1 week)
  Blood samples will be collected to determine the AUC0-Last of enlicitide chloride.
Percent Change from Baseline of Plasma Low Density Lipoprotein (LDL-C) Concentration After Administration of Enlicitide Chloride | Baseline, Week 1
  Blood samples will be collected to determine the LDL-C of enlicitide chloride.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Altasciences Clinical Kansas, Inc. (Site 0002), Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com